CLINICAL TRIAL: NCT01643018
Title: Laparoscopic Versus Open Conservative Surgery for the Management of Cystic Echinococcosis of the Liver: Prospective, Randomized, and Controlled Clinical Trial of Efficacy and Safety
Brief Title: Laparoscopic Versus Open Surgery for the Management of Cystic Echinococcosis of the Liver
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Park Gaziantep Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Kaplan, MKaplan, Medical Park Gaziantep Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MK-001-CH
Record Dates: First submitted 2012-06-26; First posted 2012-07-17 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Echinococcosis, Hepatic; Hydatid Cyst
Keywords: cystic echinococcosis; liver cyst hydatique; treatment; surgery; laparoscopy
MeSH Terms: conditions — Echinococcosis, Hepatic; Echinococcosis | interventions — Laparoscopy; Conversion to Open Surgery; Laparotomy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- laparoscopic surgery (Experimental): -Laparoscopic surgery group describes the patients treated with laparoscopic surgery
  Interventions: Procedure: laparoscopic surgery
- Open Surgery (Active Comparator): -open surgery group describes the patients treated with traditional open surgery
  Interventions: Procedure: open surgery

INTERVENTIONS:
Procedure: laparoscopic surgery — In laparoscopy group three trocars is used. The first is 10 mm and inserted within the umbilicus for telescop, the second is 10 mm and inserted just below the xiphoid process, and third is 5 mm and inserted at the right upper quadrant of the abdomen.
  Other Names: Laparoscopy
  Arms: laparoscopic surgery
Procedure: open surgery — -open surgery group describes the patients treated with traditional open surgery. In open surgery group a right subcostal incision is used.
  Other Names: laparotomy; open
  Arms: Open Surgery

SUMMARY:
Echinococcosis in humans is a parasitic tapeworm infection, caused by a larval stage (the metacestode) of Echinococcus species. The infection can be asymptomatic or severe, causing extensive organ damage and even death of the patient.

Echinococcosis is one of the most neglected parasitic diseases and the lack of the prospective randomised studies supports this idea. Development of new drugs and other treatment modalities receives very little attention, if any. In most developed countries, Cystic Echinococcosis (CE) is an imported disease of very low incidence and prevalence and is found almost exclusively in migrants from endemic regions. In endemic regions, predominantly settings with limited resources, patient numbers are high.

The aim of the hydatid cyst treatment is the death of the parasite and consequently the cure of the disease. It has to be done with a minimal risk and maximum comfort for the patient, and always paying attention to avoid complications, secondary hydatidosis, and relapses.

There are several treatment modalities. Of them the most preferred surgical method is traditional cyst management through a laparotomy incision. Same can be done with laparoscopy. In the past 15 years significant advances in laparoscopic surgical skills and techniques combined with explosive advances in laparoscopic technology have encouraged the application of laparoscopy to the evaluation and treatment of solid organs including the liver. There are many studies about the laparoscopic treatment of liver hydatid cyst published in the literature and the feasibility of this procedure has been demonstrated by them. While the majority of them are case reports or case series, there are some relatively large series comparing open versus laparoscopic surgery published in the last decade, which all are not randomized trial.

DETAILED DESCRIPTION:
This is a multicenter, balanced randomization, double blind, active-controlled, parallel-group, non-inferiority study conducted in Turkey (4 sites).

The objective of this trial is to show there is no difference in rate of recurrence 2 years after laparoscopic as compared to open management of cystic echinococcosis of the liver, by at least M (non-inferiority margin). If PLAP/POP: denotes the cure rate in the laparoscopy group (LAP) / open group (OP), then the following two-sided test problem is assessed:

H0: POP - PLAP >= M (Open Surgery is superior to Laparoscopic surgery) H1: POP - PLAP < M (Laparoscopic surgery is not inferior to open surgery)

ELIGIBILITY:
Inclusion Criteria:

* patients eighteen year-old or older
* patients diagnosed as cystic echinococcosis of the liver
* cyst number less then 3
* cyst size greater than 3 cm

Exclusion Criteria:

* previous liver surgery
* recurrent disease
* hydatid cyst with multi-organ involvement
* liver hydatid cyst complicated with infection
* contraindication for general anesthesia
* contraindication for laparoscopic surgery
* patient younger than 18
* allergy to albendazole

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2006-11; Primary Completion 2010-11 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
cyst recurrence | 24 months

SECONDARY OUTCOMES:
mortality | 24 months
intraoperative complications | 24 hours
late complications | 24 months
pain score | Post opertaive 6th hour, 1, 2, and 7th days
  VAS scoring scale will be use
patient comfort/satisfaction | 24 months
  will be measured in all follow-up examinations using a scale from 0 (worst) to 10 (excellent).
hospital stay | 10 days
  postoperative hospital days
duration of the operation | 240 minutes
  from incision to closure of the skin
quality of life | first week, 1, 6, 12, and 24 month after operation

CONTACTS AND LOCATIONS:
Overall Officials: MEHMET KAPLAN, MD, Principal Investigator — Medical Park Gaziantep Hospital, Gaziantep, Turkey
Locations (4):
- Turkey (Türkiye) (4):
  - Hatem Hospital, Gaziantep
  - Medical Park Gaziantep Hospital, Gaziantep
  - 25 Aralık State Hospital, Gaziantep
  - Dr.Ersin Aslan State Hospital, Gaziantep